CLINICAL TRIAL: NCT00943163
Title: Evaluation of Position-induced Cyclorotation Between Wavefront Measurement and Refractive Surgery by the Iris Registration Method
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 200906095R
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Eye Cyclorotation Degree; Pupil Shift
Keywords: cyclorotation; pupil; laser refractive surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cyclorotation of eyes may be affected by motion and orientation of the head and body. An automated alignment method with the technique of iris recognition was used to assess the amount and orientation of position-induced cyclorotation between preoperative wavefront measurement and laser refractive surgery.

DETAILED DESCRIPTION:
Ninety-three consecutive patients undergoing bilateral wavefront-guided laser refractive surgery in the Department of Ophthalmology of the National Taiwan University Hospital between September 2004 and December 2007 were enrolled in this retrospective study. Before laser refractive surgery, all patients were seated in front of the Zyoptix 100 system platform (Bausch & Lomb, salt lake city, UT, USA) and received Zywave aberrometer measurement on both eyes. When patients were in the supine position for refractive surgery, an infrared camera mounted on the laser system (Technolas 217z100 excimer laser system, Bausch & Lomb)obtained iris images on undilated pupils before laser ablation. Overall cyclorotation was detected by a comparison between iris images of undilated pupils in the supine position and dilated pupils in the seated position before laser treatment. The degree and direction of position-induced cyclorotation were assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing bilateral wavefront-guided laser refractive surgery

Exclusion Criteria:

* patients with strabismus, extraocular muscle palsy, muscle restriction or other diseases interfering normal ocular movement.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ninety-three consecutive patients undergoing bilateral wavefront-guided laser refractive surgery in the Department of Ophthalmology of the National Taiwan University Hospital between September 2004 and December 2007.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chih Hou, MD, Study Director — Telephone: 886-2-23123456 Ext. 65025 Email: ychou51@ntu.edu.tw
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan